CLINICAL TRIAL: NCT01211912
Title: Acetaminophen Transfer Across the Placenta and the Assessment of Fetal Well-being
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian C. Brost, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-003283
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Fetal Testing; Transplacental Transfer of Acetaminophen
Keywords: Fetal movement; Fetal breathing; Acetaminophen
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (20 patients) (Experimental): Pregnant women will be given a single dose of 1000 mg of acetaminophen orally after a baseline ultrasound and 60 minutes before a repeat ultrasound.
  Interventions: Drug: Arm 1 (20 patients)
- Arm 2 (34 patients) (Experimental): Pregnant women will be given a single dose of 1000 mg of acetaminophen orally 30 minutes to 24 hours before a scheduled cesarean section.
  Interventions: Drug: Arm 2 (34 patients)

INTERVENTIONS:
Drug: Arm 1 (20 patients) — Acetaminophen 1000 mg by mouth once
  Other Names: Tylenol
  Arms: Arm 1 (20 patients)
Drug: Arm 2 (34 patients) — Acetaminophen 1000 mg by mouth once
  Other Names: Tylenol
  Arms: Arm 2 (34 patients)

SUMMARY:
This study has two aims:

1. to evaluate placental transfer of acetaminophen from mother to baby transplacentally given from 30 minutes to 24 hours prior to cesarean delivery (34 patients)
2. to understand the impact of maternal acetaminophen use on fetal movement and breathing (20 patients)

ELIGIBILITY:
Inclusion Criteria

* Pregnant females
* Age 18-44
* Any race
* Any parity
* Singleton Gestations
* Weight between 60-90 kg

Exclusion Criteria

* Acetaminophen Allergy
* Contraindication to Acetaminophen Use
* Chorioamnionitis
* Preeclampsia
* Diabetes Mellitus
* Placental Abruption
* Placenta Previa
* Fetal Anomaly
* Intrauterine growth restriction (IUGR)
* Multiple Gestations
* Maternal Medical Disease
* Acetaminophen use in the last 3 days
* Plan to donate or bank fetal cord blood

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maternal and neonatal serum acetaminophen level | Time Frame: 30 minutes to 24 hours post administration
  Pregnant women will be given 1000 mg of acetaminophen orally and have both maternal and neonatal serum acetaminophen levels checked at the time of cesarean section 30 minutes to 24 hours after administration.
Fetal breathing and body movements | Time Frame: 60 minutes
  Pregnant women will have a baseline assessment of fetal breathing and body movements with ultrasound and will then be given 1000 mg of acetaminophen orally. Fetal breathing and body movements will then be reassessed 60 minutes later.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Brost, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States